CLINICAL TRIAL: NCT06465303
Title: An Exploratory, Randomised, Double-blind, Multicentre, Placebo-controlled Study of RTP-026 to Assess Safety, Tolerability and Efficacy in Patients With ST-Elevation Myocardial Infarction (STEMI)
Brief Title: A Study of RTP-026 to Assess Safety, Tolerability and Efficacy in Patients With ST-Elevation Myocardial Infarction (STEMI)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: ResoTher Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ResoTher-CS002
Record Dates: First submitted 2024-06-13; First posted 2024-06-18 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: ST Elevation Myocardial Infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- RTP-026 (Experimental)
  Interventions: Drug: RTP-026
- Placebo (Experimental)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RTP-026 — Intervention is for each subject administered as three 30-minutes infusions of either A: 25μg/kg RTP-026; or B: ≥ 26μg/kg and ≤75μg/kg RTP-026; or C: A maximum of 3 x treatment dose RTP-026 as given in B;
  Arms: RTP-026
Drug: Placebo — Intervention is for each subject administered as three 30-minutes infusions of placebo
  Arms: Placebo

SUMMARY:
This is an exploratory, randomized, double-blind, multicentre, placebo-controlled study of RTP-026.

The study population will consist of men and women with documented evidence of ST-elevation myocardial infarction (STEMI) referred to primary Percutaneous Coronary Intervention (PCI).

DETAILED DESCRIPTION:
An exploratory, randomized, double-blind, multicentre, placebo-controlled study of RTP-026 to assess safety, tolerability, and efficacy in patients with (STEMI).

The study population is men between 18-85 years and post-menopausal women up to 85 years with documented evidence of STEMI referred to primary PCI with acute onset of chest pain lasting <12 hours and neutrophil to lymphocyte ratio (NLR) in the range of 3-17 at hospital admission (Please refer to inclusion criteria).

The participants will be given three 30-minute intravenous infusions of RTP-026 or placebo (the investigational product). The first dose is to be initiated within 2 hours following the establishment of reflow after PCI, and the following two study treatments with 8-hour intervals.

The purpose of this study is to evaluate the safety, tolerability and efficacy of RTP-026 versus placebo in multiple doses.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent for participation in the study has been obtained prior to initiating any study-specific procedures
* Men between 18-85 years of age and post-menopausal women up to 85 years of age
* Acute onset of chest pain of < 12 hours duration
* STEMI as characterized on ECG by 2 mm ST elevation in 2 or more V1 through V4 leads or presumed new left bundle branch block with a minimum of 1 mm concordant ST elevation or 1 mV ST elevation in the limb lead (II, III and aVF, I, aVL) and V4-V6 or ST depression in 2 or more V1 through V4 leads indicating posterior acute myocardial infarction (AMI)
* Eligible for primary PCI
* NLR in the range of 7-17 at hospital admission. In patients with chest pain lasting > 3 - ≤ 6 hours at admission, the NLR should be in the range of 4.8-17 and for patients with chest pain lasting ≤ 3 hours at admission, the NLR should be in the range of 4.8-17, or the neutrophile count should be ≥ 9 x 10E9/L, irrespective of the lymphocyte count. For STEMI patients with an anterior or anterolateral infarction, the NLR should be ≥3.

Exclusion Criteria:

* Participation in any other study involving investigational drug(s) during the study and within 4 weeks prior to study entry
* Previous exposure to RTP-026
* Time from symptoms onset to primary PCI > 12 hours
* Previous CABG
* Evidence of active malignant disease
* Ongoing treatment with immune suppressive compounds
* Any condition that, in the view of the investigator, would suggest that the patient is unable to comply with the study protocol and procedures
* Known contraindications to CMR
* ORBI Risk Score > 12

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2024-07-16 (Actual); Primary Completion 2025-12-21 (Estimated); Study Completion 2025-12-21 (Estimated)

PRIMARY OUTCOMES:
Change in Cardiac Troponin T (cTNT) | 24 hours
  Change in cTnT determined in blood samples taken at Baseline, 6 hours post-PCI, before the infusion 3 and 24 hours post-PCI.
Change in Creatinine kinase-MB (CK-MB) | 24 hours
  Change in CK-MB determined in blood samples taken at Baseline, 6 hours post-PCI, before the infusion 3 and 24 hours post-PCI.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Engstrøm, Prof. MD, Principal Investigator — Hjertecenteret, Rigshospitalet, Denmark
Locations (1):
- Hjertecenteret, Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No